CLINICAL TRIAL: NCT04906564
Title: RNF213 Variants and Collateral Vessels in Moyamoya Disease
Status: Completed | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY 2017-141-01
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Moyamoya Disease
Keywords: Moyamoya Disease; RNF213 Variants; Collateral Vessels
MeSH Terms: conditions — Moyamoya Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Moyamoya disease patients: Moyamoya disease patients' inclusion Criteria:
  1. Written informed consent is obtained; 2. Patients with age between 4-60 years; 3. Cerebral digital subtraction contrast angiography (DSA) reveal severe stenosis or occlusion of the distal internal carotid or proximal middle and anterior cerebral arteries with prominent lenticulostriate 'moyamoya collaterals'.
  Exclusion Criteria:
  1. There are other vascular diseases, including systemic vasculitis, neurofibroma, meningitis, sickle cell disease, down's syndrome, and previous basilar radiotherapy; 2. Patients with cardiogenic embolism, including a history of atrial fibrillation, valvular disease or cardiac valve replacement; 3. Physical or subjective failure to cooperate with the examination or serious comorbid diseases.
  Interventions: Other: Identification of genetic variants

INTERVENTIONS:
Other: Identification of genetic variants — Identification of genetic variants

SUMMARY:
The purpose of this study is to detect the association between RNF213 variants and collateral vessels in patients with moyamoya disease.

DETAILED DESCRIPTION:
Moyamoya disease (MMD) is a chronic cerebrovascular disorder characterized by the presence of occlusion which occurs at the internal carotid arteries and their main branches during the development of a basal collateral network. The ring finger 213 (RNF213) was identified as a strong susceptibility gene in patients with MMD in East Asia. The role of RNF213 variants in pathogenesis of MMD is still unclear. Specific "moyamoya vessels" correlate with the onset of stroke. The purpose of this study is to investigate the relationship between RNF213 variants and collateral vessels in patients with moyamoya disease, and provide potential pathogenesis of moyamoya disease.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained
* Patients with age between 4-60 years
* Cerebral digital subtraction contrast angiography (DSA) reveal severe stenosis or occlusion of the distal internal carotid or proximal middle and anterior cerebral arteries with prominent lenticulostriate 'moyamoya collaterals'

Exclusion Criteria:

* There are other vascular diseases, including systemic vasculitis, neurofibroma, meningitis, sickle cell disease, down's syndrome, and previous basilar radiotherapy
* Patients with cardiogenic embolism, including a history of atrial fibrillation, valvular disease or cardiac valve replacement
* Physical or subjective failure to cooperate with the examination or serious comorbid diseases

Ages: 4 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Moyamoya disease patients
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Identification of RNF213 variants and different types of collateral vessels | Baseline

SECONDARY OUTCOMES:
Identification of serum biomarkers and different types of collateral vessels | Baseline
  Hcy, HDL, LDL, ApoA, ApoB et al.
Identification of clinical characteristics and different types of collateral vessels | Baseline
  Age, Gender, Clinical manifestations, Comorbidities, BMI et al.
Identification of RNF213 variants, serum biomarkers, clinical characteristics and different types of postoperative collateral vessels | 6-12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No